CLINICAL TRIAL: NCT07392086
Title: Comparison of the Effects of Flow-Controlled Ventilation (FCV) and Volume-Controlled Ventilation (VCV) on Respiratory Mechanics and Gas Exchange During One-Lung Ventilation: A Multicenter Prospective Observational Study (FCVOLVent)
Brief Title: Comparison of FCV and VCV in One-Lung Ventilation
Acronym: FCVOLVent
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Collaborators: Kocaeli City Hospital (Other Government); Yedikule Training and Research Hospital (Other); Sakarya University (Other); Ataturk University (Other)
Responsible Party: Principal Investigator, Hakan Miniksar, Associate Professor of Anesthesiology and Reanimation, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-11/1250
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: One-lung Ventilation (OLV); Thoracic Surgery; Respiratory Mechanics
Keywords: Flow-Controlled Ventilation; Thoracic Anesthesia; Volume-Controlled Ventilation; One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All participants: One-Lung Ventilation with Volume-Controlled Ventilation (VCV)
- Prospective observational cohort study: Flow-Controlled Ventilation during One-Lung Ventilation

SUMMARY:
One-lung ventilation (OLV) is commonly used during thoracic surgery but may negatively affect lung mechanics and gas exchange. Different ventilation strategies are used during OLV, and their effects on respiratory parameters remain an important clinical concern.

Flow-controlled ventilation (FCV) is a newer ventilation mode that allows precise control of inspiratory and expiratory flow, potentially improving lung mechanics and gas exchange. Volume-controlled ventilation (VCV) is a widely used conventional ventilation strategy during thoracic anesthesia.

The FCVOLVent study is a multicenter, prospective observational study designed to compare the effects of FCV and VCV during one-lung ventilation in adult patients undergoing thoracic surgery. Patients will be ventilated with either FCV or VCV as part of routine clinical practice.

The study aims to evaluate respiratory mechanics and oxygenation parameters, including the PaO₂/FiO₂ ratio, airway pressures, lung compliance, and mechanical power during surgery. Data will be collected at predefined time points during one-lung ventilation.

The results of this study are expected to provide real-world clinical evidence on the potential advantages and limitations of flow-controlled ventilation compared with volume-controlled ventilation during one-lung ventilation.

DETAILED DESCRIPTION:
Detailed Description

One-lung ventilation (OLV) is a fundamental anesthetic technique in thoracic surgery; however, it is frequently associated with impaired respiratory mechanics, ventilation-perfusion mismatch, and compromised gas exchange. Volume-controlled ventilation (VCV) is the most commonly used ventilation mode during OLV, but it may result in uneven gas distribution, higher peak airway pressures, and potential lung injury.

Flow-controlled ventilation (FCV) is a novel ventilation mode characterized by constant and controlled inspiratory and expiratory flow, allowing precise regulation of airway pressures and lung volumes. Previous experimental and limited clinical data suggest that FCV may improve lung recruitment, optimize respiratory mechanics, and enhance gas exchange compared with conventional ventilation strategies.

The FCVOLVent study is a multicenter, prospective observational study designed to compare the effects of FCV and VCV on respiratory mechanics and gas exchange in adult patients undergoing thoracic surgery requiring one-lung ventilation. Patients will be ventilated according to the ventilation strategy routinely used at each participating center, either FCV or VCV, without randomization or intervention beyond standard clinical practice.

Primary outcomes include intraoperative respiratory mechanics parameters such as dynamic compliance, airway pressures, and driving pressure during OLV. Secondary outcomes include arterial blood gas variables, oxygenation indices, carbon dioxide elimination, and selected perioperative clinical parameters.

Data will be collected at predefined time points during two-lung ventilation and one-lung ventilation phases. The study aims to provide real-world clinical evidence regarding the potential advantages and limitations of FCV compared with VCV in thoracic anesthesia practice.

By evaluating ventilation strategies across multiple centers, the FCVOLVent study seeks to contribute to a better understanding of lung-protective ventilation approaches during one-lung ventilation and to inform future interventional trials in this field.

ELIGIBILITY:
Inclusion Criteria Adult patients aged 18 years and older Patients undergoing thoracic surgery requiring one-lung ventilation (OLV) Requirement for one-lung ventilation for at least 30 minutes American Society of Anesthesiologists (ASA) physical status I-III Provision of written informed consent Patients ventilated with flow-controlled ventilation (FCV) or volume-controlled ventilation (VCV) as part of routine clinical practice

Exclusion Criteria Requirement for emergency surgery History of untreated asthma High pulmonary risk, defined as predicted postoperative FEV₁ < 20 mL/kg in males and < 18 mL/kg in females High cardiac risk, including advanced cardiomyopathy with left ventricular ejection fraction < 30% Body mass index (BMI) > 35 kg/m² Contraindication to total intravenous anesthesia (TIVA) Evidence of pulmonary infection prior to surgery Presence of other significant pulmonary pathologies (e.g., tuberculosis, bullous lung disease, bronchiectasis) Severe COPD (GOLD stage III-IV) or significant restrictive lung disease Age < 18 years or > 80 years, or pregnancy ASA physical status IV or higher Uncontrolled arrhythmia or history of myocardial infarction within the past 3 months Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older undergoing thoracic surgery requiring one-lung ventilation with flow-controlled ventilation (FCV) or volume-controlled ventilation (VCV).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Capacity | Intraoperative period (during one-lung ventilation)
  PaO₂/FiO₂ Ratio

SECONDARY OUTCOMES:
Respiratory parameters | Intraoperative period (during one-lung ventilation)
  mechanical power (MP)

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Miniksar, Study Chair — Health Sciences University Dr. Abdurrahman Yurtarslan Ankara Oncology Training and Research Hospital
Locations (1):
- Health Sciences University Dr. Abdurrahman Yurtarslan Ankara Oncology Training and Research Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bialka S, Palaczynski P, Szuldrzynski K, Wichary P, Kowalski D, van der Hoorn JWA, Bottinger L, Misiolek H. Flow-controlled ventilation - a new and promising method of ventilation presented with a review of the literature. Anaesthesiol Intensive Ther. 2022;54(1):62-70. doi: 10.5114/ait.2022.112889. PMID 35142160